CLINICAL TRIAL: NCT05909085
Title: A Randomized Double Blinded Controlled Trial to Investigate the Impact of Needle Manipulation and Accuracy of Between Two Commercially Available Ultrasound Devices
Brief Title: The Impact of Needle Manipulation and Accuracy Between Hand Held Automatic and Traditional Ultrasound Device
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2000034863; No NIH funding 09.05.23 (Other: Yale)
Record Dates: First submitted 2023-06-01; First posted 2023-06-18 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Labor Analgesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Handheld traditional ultrasound (Active Comparator): Traditional US will be used to compare number of needle manipulations to the handheld US.
  Interventions: Device: Traditional ultrasound
- Handheld Automated ultrasound (Other): Automated device provides automatic information pertaining to distance to epidural space distance and interspace location.
  Interventions: Device: Automated ultrasound

INTERVENTIONS:
Device: Traditional ultrasound — Labor epidural will be performed after marking patient skin using traditional ultrasound guidance
  Arms: Handheld traditional ultrasound
Device: Automated ultrasound — Labor epidural will be performed after marking patient skin using an automated ultrasound device
  Arms: Handheld Automated ultrasound

SUMMARY:
In this double blinded randomized controlled trial, the investigators would like to compare the effects on needle manipulation when relatively inexperienced sonographist (< 1 year of ultrasound experience) perform ultrasound guided labor epidurals utilizing a traditional handheld ultrasound versus a handheld device that was engineered to provide automated guidance. The primary outcome of this study would be number of needle passes.

DETAILED DESCRIPTION:
Patient will be approached upon admission to labor and delivery floor (Standard of care). The study will be presented to the patient and if they agree, they will be consented. (Study). Upon epidural patient request patient will be randomized to A-US vs B-US based on the randomization table. Ten envelopes will be available with the randomization choice. (Study). The resident will walk in with both US devices into the room (for patient blinding) and perform scan with the device the randomization table called for. (Study). After performing scan and markings of the patients back, the research fellow or clinical fellow will be called into the room to evaluate the number of needle manipulation and provide surveys related to patient and labor analgesia satisfaction. (Study).

Number of needle insertion attempts: defined as advancement of the needle through the skin in an effort to enter the epidural space; a needle requiring withdrawal from the skin for reinsertion is to be counted as an additional insertion attempt. Time to landmark identification: defined as the time interval between the start of needle puncture site identification and the time to first needle puncture attempt. The start time of needle puncture site identification in both the LT and UST corresponds to when the resident physician first places his/her hand on the patient to palpate the back. In both groups, all materials, supplies, and equipment will be prepared and readily available prior to the start of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* ASA-1, ASA-2, and ASA-3
* Patients with no known back deformities
* Ability to sit upright for epidural placement
* No prior lumbar surgery
* No allergies to ultrasound gel

Exclusion Criteria:

* Coagulopathy
* Low platelet count
* Allergies to local anesthetics

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of needle passes | From local anesthetic injection (time 0) till Loss of resistance (in minutes), up to 60 minutes
  Number of ventral needle movements without removing needle from skin. A needle pass is defined as any forward advancement or withdraw and forward redirection of the needle without withdraw from the skin.

SECONDARY OUTCOMES:
Number of Needle attempts | From local anesthetic injection (time 0) till Loss of resistance (in minutes), up to 60 minutes
  Number of times the needle is advanced in and out of the skin
Time to obtain ultrasound images with traditional ultrasound device | Time at which ultrasound device is placed on patients back (time 0) until image obtained (in minutes), up to 30 minutes
  Time from placing ultrasound on patients back until markings are complete
Time to obtain images with automated ultrasound device | Time at which ultrasound device is placed on patients back (time 0) until image obtained (in minutes), up to 30 minutes
  Time from placing ultrasound on patients back until markings are complete
Time from local anesthetic injection till time of epidural space identification | Up to 60 minutes
  Time will be recorded once local anesthetic is injected and stopped upon obtaining loss of resistance
Accuracy of handheld ultrasound - difference between predicted epidural space distance minus actual needle distance | Up to 60 minutes
  Accuracy will equal the difference between the estimated depth calculated by the device - actual needle depth as measured from skin to epidural space in centimeters.
Accuracy of automated ultrasound device - difference between predicted epidural space distance minus actual needle distance | Up to 60 minutes
  Accuracy will equal the difference between the estimated depth calculated by the device - actual needle depth as measured from skin to epidural space in centimeters.
Patient satisfaction | 15 - 20 minutes after epidural placement
  Assessed after the administration of the loading dose. Patient will be asked to rate their pain on a scale 0-10, 0 = not satisfied, 10 = completely satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gonzalez, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vallejo MC, Phelps AL, Singh S, Orebaugh SL, Sah N. Ultrasound decreases the failed labor epidural rate in resident trainees. Int J Obstet Anesth. 2010 Oct;19(4):373-8. doi: 10.1016/j.ijoa.2010.04.002. Epub 2010 Aug 8. PMID 20696564
- [Result] Carvalho B, Seligman KM, Weiniger CF. The comparative accuracy of a handheld and console ultrasound device for neuraxial depth and landmark assessment. Int J Obstet Anesth. 2019 Aug;39:68-73. doi: 10.1016/j.ijoa.2019.01.004. Epub 2019 Jan 11. PMID 30770208
- [Result] Weiniger CF, Carvalho B, Ronel I, Greenberger C, Aptekman B, Almog O, Kagan G, Shalev S. A randomized trial to investigate needle redirections/re-insertions using a handheld ultrasound device versus traditional palpation for spinal anesthesia in obese women undergoing cesarean delivery. Int J Obstet Anesth. 2022 Feb;49:103229. doi: 10.1016/j.ijoa.2021.103229. Epub 2021 Sep 23. PMID 34670725
- [Result] Seligman KM, Weiniger CF, Carvalho B. The Accuracy of a Handheld Ultrasound Device for Neuraxial Depth and Landmark Assessment: A Prospective Cohort Trial. Anesth Analg. 2018 Jun;126(6):1995-1998. doi: 10.1213/ANE.0000000000002407. PMID 28858898